CLINICAL TRIAL: NCT06547762
Title: Hybrid Approach (In-person and Remote) to Pediatric Rehabilitation: A Look Beyond the Corona Crisis 2019
Brief Title: Hybrid Approach to Pediatric Rehabilitation
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Alyn Pediatric & Adolescent Rehabilitation Hospital (Other)
Collaborators: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Naomi Gefen, PI, PARC ALYN; Deputy Director General, Alyn Pediatric & Adolescent Rehabilitation Hospital
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 063-22
Record Dates: First submitted 2024-07-17; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Cerebral Palsy; Traumatic Brain Injury; Orthopedic Disorder
Keywords: Occupational Therapy; Physical Therapy; Speech and Language Pathology; Psychology; Telerehabilitation; Hybrid Rehabilitation
MeSH Terms: conditions — Cerebral Palsy; Brain Injuries, Traumatic; Musculoskeletal Diseases; Speech

STUDY DESIGN:
Intervention Model Description: Control group and Intervention group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hybrid rehabilitation (Experimental): Children will receive one day of remote rehabilitation. All other days children will receive therapy at hospital
  Interventions: Other: Hybrid approach (in-person and remote) to pediatric rehabilitation: A look beyond the COVID-19 crisis

INTERVENTIONS:
Other: Hybrid approach (in-person and remote) to pediatric rehabilitation: A look beyond the COVID-19 crisis — Hybrid rehabilitation. Out patients will receive one day a week of remote therapy and the remaining (1-4 days) in person at rehabilitation hospital

SUMMARY:
Children and youth recovering from acquired injuries typically receive therapy via in-patient or outpatient rehabilitation (OPR). Families from peripheral areas often face significant time and financial burdens to access treatment. Over the past decade, evidence supporting the effectiveness of remote (online) rehabilitation has increased.

Objectives: 1. Identify facilitators and barriers to hybrid service adoption. 2. Develop a hybrid telerehabilitation program for youth that is at least equivalent (non-inferior) to conventional, in-person therapy. 3. Compare hybrid rehabilitation to in-person rehabilitation at two centers in Israel in terms of: Adherence to therapy, Therapeutic alliance, Perceived quality of care (families and therapists), Functional effectiveness (measured by pre-post change in the Pediatric Evaluation of Disability Inventory, PEDI), Cost-effectiveness (including training requirements, physical space requirements, and costs); 4. Provide best practice recommendations for hybrid rehabilitation in children.

Research Methods: Focus Groups: Experts will develop a two-month hybrid program for approximately 200 children in OPR, commencing one month after in-person rehabilitation.

Evaluation Metrics: Therapy adherence, therapeutic alliance, and perceived quality of care will be assessed monthly and compared to in-person treatment. Insights will inform best practice guidelines for hybrid telerehabilitation.

Data Collection: Thematic Analysis: Analyzing focus group information. Comparative Metrics: Comparing measures of adherence, therapeutic alliance, and perceived quality of care between hybrid and in-person programs.

Difference-in-Difference Approach: Assessing functional differences between in-person and remote therapy.

Cost Analysis: Estimating direct and indirect costs per child for in-person versus remote rehabilitation.

DETAILED DESCRIPTION:
Scientific background: Children and youth recovering from acquired injuries receive therapy via in-patient or outpatient rehabilitation (OPR). Families from the periphery are required to invest time and money to get treatment. In the last decade, evidence for the effectiveness of remote (online) rehabilitation has grown. During the first four months of the COVID-19 pandemic, remote rehabilitation services were provided at Sheba and Alyn Medical Centers with demonstrated feasibility and satisfaction. Nevertheless, most rehabilitation services returned to in-person treatment. Objectives: To develop, implement and evaluate hybrid OPR for youth including a) identification of facilitators and barriers to hybrid service adoption; b) development of a hybrid telerehabilitation program for youth that is at least equivalent (non-inferior) to conventional, in-person therapy; c) compare hybrid rehabilitation to in-person rehabilitation at two rehabilitation centers in Israel in terms of (1) adherence to therapy, (2) therapeutic alliance and (3) perceived quality of care (families and therapists), (4) functional effectiveness as measured by pre-post change in the PEDI, (5) cost-effectiveness of hybrid therapy (by comparing financial versus effectiveness outcomes) in the healthcare system (hospitals, health maintenance organizations), including training requirements, physical space requirements and cost. d) provide best practice recommendations for hybrid rehabilitation in children.

Working hypotheses: 1) Carrying out research at two major rehabilitation centers will enable identification of target populations for hybrid rehabilitation programs, assessment of the required resources and provision of solutions to identified barriers; 2) families and caregivers will express positive attitudes toward hybrid rehabilitation.3) the hybrid program will be cost-effective in terms of direct and indirect costs.

Research Methods: Focus groups of experts will develop a two-month hybrid program offered to all children (~200) in OPR commencing one month after in-person rehabilitation. Therapy adherence, therapeutic alliance and perceived quality of care will be examined monthly and compared to in-person treatment. Insight will be used to formulate best practice guidelines for hybrid telerehabilitation.

Data Collection: Thematic analysis will be used to analyze focus groups information. Data on measures of adherence, therapeutic alliance and perceived quality of care will be compared between hybrid and in-person programs. A difference-in-difference approach will assess differences in function between in-person and remote therapy. Cost estimates will compare direct and indirect services per child for in-person versus remote rehabilitation.

Importance of research: This study will be among the first to examine implementation of a hybrid program as recommended by the Ministry of Health (MOH) 'Remote Medicine' (6/2019, section 4.4). Utilizing the demonstrated benefits and infrastructure developed for remote rehabilitation during Corona pandemic , this research will help to uphold a basic principle in the State Health Insurance Law - ensuring accessible and quality health services throughout the country.

Possible recommendations for policy makers: Best practices for hybrid rehabilitation programs will enable policy makers to make quality rehabilitation services more accessible nationwide.

ELIGIBILITY:
Inclusion Criteria:

* Children with physical disability
* Children receiving treatment via the out patient department
* Children who receive more than one day of treatment a week.
* Children who are able to follow instructions
* Families who can interact with a computer and other technologies

Exclusion Criteria:

* Children who are visually impaired
* Children who are hearing impaired
* Children who receive hydrotherapy every day of their rehabilitation program

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-08-16 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Adherence to therapy | 2 months
  Each child is prescribed a rehabilitation program. This outcome will follow the number of times that the child participated in the sessions- comparing to the prescribed program. For example if the child was supposed to participate in 5 weekly sessions and only participated in 3 sessions. The ratio of number of treatments performed to the number prescribed=adherence. A higher value indicates ahigher adherence level.
Therapeutic alliance | 2 months
  We will use the Working Alliance Inventory (WAI) (Horvath & Greenberg, 1989), a self-report questionnaire designed to assess the structure of the therapeutic alliance. The items are rated on a 7-point scale (never to always). A higher scores reflect a higher quality of therapeutic alliance.
Perceived quality of care- therapists | 2 months
  The Clinician Evaluation of Tele rehabilitation Service (CETS) (Krasovsky et al., 2021) questionnaire for evaluating clinicians' feedback on tele rehabilitation will be completed. The scale is 1-5, with the higher score being better.
Perceived quality of care- families | 2 months
  For families the System Usability Scale (SUS) will be used, it is a10 item 5-point Likert scale to assess the user experience and perception of quality of care of the hybrid and in-person programs (Brooke, 1996). A higher score is better
Cost-effectiveness of hybrid therapy | 2 months
  We will assess direct costs of in-person services, including direct payment schedules per week, for each treatment modality. Additionally, we will ask parents to complete information on travel (time and costs) and related expenses. The costs will be reported in monetary units

SECONDARY OUTCOMES:
Improved Function | 2 months
  The child's function will be assessed by the using the Pediatric Evaluation of Disability Inventory (PEDI). The Hebrew PEDI will be used (Elad et al., 2012).
  The PEDI is a valid and reliable measure of basic activities of daily living. The scores are on a scale of 0-3, with a higher score indicating higher function.

CONTACTS AND LOCATIONS:
Locations (1):
- Alyn Pediatric and Adolescent Rehabilitation Center, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No